CLINICAL TRIAL: NCT05601050
Title: Linguistic Predictors of Outcomes in Psychosis
Acronym: LPOP
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Winterlight Labs (Industry)
Responsible Party: Principal Investigator, Sunny Tang, Assistant Professor, Northwell Health
Other Study IDs: 20-0460
Record Dates: First submitted 2022-10-25; First posted 2022-11-01 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia and Related Disorders
Keywords: Schizophrenia; speech; language; language processing; digital health
MeSH Terms: conditions — Schizophrenia; Speech; Language

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PSD (Psychosis spectrum disorder) group: Current DSM-V-defined diagnosis of schizophrenia, schizophreniform, schizoaffective disorder, unspecified psychotic disorder, or brief psychotic disorder, or bipolar 1 disorder with psychotic features or major depressive disorder with psychotic features using the Structured Clinical Interview for Axis I DSM-V Disorders (SCID-I/P).
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
Longitudinal observational study of the relationship between speech patterns and clinical symptoms in schizophrenia spectrum disorders.

DETAILED DESCRIPTION:
The accurate prediction and tracking of clinical and functional outcomes in young people with schizophrenia-spectrum disorders is critical for delivering appropriate interventions and for understanding the brain mechanisms behind psychosis. Language is an optimal avenue for tracking psychosis processes because language is readily produced and captured, has well-established disruptions in psychosis, and known relationship to brain circuits. Using computers to automate detection of language features has the further advantage of being objective, quantitative, and adaptable into an efficient and cost-effective tool. The investigators propose to use automated linguistic analyses in young people early in the course of schizophrenia spectrum disorders to measure language features including fluency (speech rate), complexity (proportion of unique words), prosody (changes in tone during speech), and semantic coherence (how sequencing of words conform to expected patterns).

The investigators will test whether these features meaningfully reflect clinical symptoms, cognition, and functioning, and whether they help predict how psychosis symptoms change over time.

ELIGIBILITY:
Inclusion Criteria:

* Speaks English with conversational proficiency
* Current DSM-V-defined diagnosis of schizophrenia, schizophreniform, schizoaffective disorder, unspecified psychotic disorder, or brief psychotic disorder or bipolar 1 disorder with psychotic features or major depressive disorder with psychotic features using the Structured Clinical Interview for Axis I DSM-V Disorders (SCID-I/P).
* Current significant positive or disorganized symptoms of psychosis (DSM 5 Criterion A) including rating at or above any of the following on the BPRS:
* Grandiosity (Severe - 6)
* Suspiciousness (Moderately Severe - 5)
* Hallucinations (Moderately Severe - 5)
* Unusual thought content (Moderate - 4)
* Bizarre Behavior (Moderate - 4)
* Disorientation (Moderate - 4)
* Conceptual Disorganization (Moderate - 4)
* Early phase of psychotic illness as defined by less than 2 years elapsed since reaching threshold for psychotic disorder
* Age 15 to 40 years
* Has capacity and willing to sign informed consent; if minor, parent is willing to give consent and child is willing to give assent.
* Screening will not include a pregnancy test. Pregnant women will not be screened out of the study because the study procedures are of very low risk overall, and pregnancy does not place the participant or the fetus at any significant risk.
* Minors will be included in the study because psychosis symptoms frequently onset before the age of 18 and this patient group is particularly in need of accurate prognosis and treatment. Therefore, it is of vital importance that the conclusions of the study be applicable to minors and that they be included among the participants.

Exclusion Criteria:

* Participants with substance-induced psychotic disorder, a psychotic disorder due to a general medical condition, delusional disorder, or shared psychotic disorder will not be included.
* Patient currently under the influence of alcohol or drugs.
* Disorders affecting speech or language, such as aphasia, intellectual disability (IQ<70), or language disorder, or movement disorders affecting speech like tardive dyskinesia, or physical impairments causing significant distortions to speech
* Serious neurological or endocrine disorder or any medical condition or treatment known to affect the brain and/or language, including but not limited to: neurodegenerative disorders, traumatic brain injury with active symptoms, autism spectrum disorder, encephalitis, epilepsy
* Significant risk of suicidal or homicidal behavior;
* Cognitive or language limitations, or any other factor that would preclude subjects providing informed consent

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Inpatients will be recruited from Northwell Health. Patients whose treatment team believes they would be appropriate for a research study will be approached by research staff and the research project will be explained to them in detail. Potential participants will also be screened for by reviewing newly admitted patients to the inpatient units. Educational seminars regarding this study may be held to inform clinicians and staff of our goals and protocol. Potential participants will be made aware that declining participation will not affect their care.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Speech features from the Winterlight Speech Assessment | 6 months
  Acoustic and linguistic measures of speech computed based on performance on the Winterlight Speech Assessment.

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) | 6 months
  18 item, range = 1, not observed - 7, very severe; higher scores resulting in worse outcome.
Hamilton Rating Scale for Depression | 6 months
  24 item, range = 0, absent - 4, severe; higher scores resulting in worse outcome.
Young Mania Rating Scale | 6 months
  11 item, range = 0, absent - 8, severe; higher scores resulting in worse outcome.
Scale for the Assessment of Negative Symptoms | 6 months
  22 item, range= 0, absent - 5, severe; higher scores resulting in worse outcome.
Scale for the Assessment of Thought Language and Communication | 6 month
  20 item, range= 0, absent - 3, severe; higher scores resulting in worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sunny X Tang, MD, Principal Investigator — Northwell Health, The Feinstein Institutes of Medical Research
Locations (1):
- Zucker Hillside Hospital, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: No